CLINICAL TRIAL: NCT04910672
Title: Effectiveness of Osteopathic Treatment in Patients With Primary Dysmenorrhea
Brief Title: Primary Dysmenorrhea and Osteopathic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Escuela de osteopatía de Madrid (Other)
Collaborators: University of Seville (Other)
Responsible Party: Principal Investigator, Sara Santiago Tello, physiotherapist, Escuela de osteopatía de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OsteopatiaMadrid; MCLozano (Other: OsteopatiaMadrid)
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Pain; Pelvic Pain Syndrome; Sexual Dysfunction
Keywords: Primary Dysmenorrhea; Spinal Manipulation; Pelvic Pain; Pain Threshold; Sexual Dysfunctions; Osteopathic Treatment; Manual therapy; Visceral Manipulation
MeSH Terms: conditions — Pelvic Pain; Sexual Dysfunction, Physiological | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This is a double-blind prospective, longitudinal, randomized, controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator does not participate in the randomization process. Participants will be blinded as to which treatment group they belong to. The experimental group will not know the treatment time, the type of treatment or the sessions received by the control group, or vice versa.
  The researcher who will carry out the pre- and post-measurements will be blinded in relation to the type of intervention.
  The investigator who will perform the statistical analysis will be blinded with respect to the type of intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group (n = 30) will only carry out a bilateral global pelvic manipulation
  Interventions: Other: Control Group
- Experimental Group (Experimental): The experimental group (n = 30) will be treated following an osteopathic treatment, through a bilateral global pelvic manipulation and a specific internal technique for mobility of the cervix
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Control Group — Bilateral global pelvic manipulation. Lower right limb in extension. The left lower limb in flexion, until the tension on the SPIS was felt. Introduce very little rotation of the spine. ASI anterior slide until crease forms at waist.
  We bring the elbow towards our hips. We rotate the patient posteriorly to open the lumbo sacral facet. The thrust is performed by simultaneously increasing these three parameters, with kick and joint compression.
  Arms: Control Group
Other: Experimental Group — Bilateral Global Pelvic Manipulation and Internal Correction Technique for Laterflexion of the Uterus The technique consists of making contact with the vaginal fingers on the upper and anterior part of the cervix, while the abdominal hand, dragging the skin towards the pubis, tries to make contact as posterior as possible on the fundus of the uterus. The technique consists, while the patient breathes widely, in progressively raising the uterine fundus forward and upward and lowering the cervix until the normal anteversion position is achieved.
  At the end of the technique, fixing the correction position of the uterus, we can ask the patient to perform a pelvic anteversion, while the correction is maintained. At the end of the technique, all abnormal tension should have disappeared and the uterus should have recovered a physiological position of anteversion.
  Arms: Experimental Group

SUMMARY:
This study is adressed to women with primary dysmenorrhea, it´s a gynecological disorder that is defined as colicky pain associated with menstruation and is located in the lower abdomen and in the lumbo-pelvic area. It appears between the first 8-72 hours and four days of the menstrual cycle and affects almost 85% of women, 30% of them severely. This study aims to demonstrate that osteopathic manual therapy is an effective therapeutic option in patients with primary dysmenorrhea. Another objective is to verify that osteopathic manual treatment provides an improvement in the intensity of pain, quality of life and a reduction in the consumption of medicines in these patients.

DETAILED DESCRIPTION:
It will be a prospective study, a double-blind randomized controlled clinical trial. The sample group will include 60 patients, between 18 and 30 years old divided into two experimental groups. The experimental group (n = 30) will be treated following an osteopathic treatment, through a bilateral global pelvic manupulation (GPM) and a specific internal technique for mobility of the cervix, and the control group (n = 30) will only carry out a bilateral GPM. A measurement will be made before the first treatment, another after each session, and the last one two weeks after the last intervention (anthropometric measurements, quality of life questionnaire, sexual health, osteopathic tests, pressure point with algometer, pain and medicines consumption). The established outcome measures are: pain intensity according to the visual analog scale (VAS), depression points measured with an algometer, a health-related quality of life questionnaire, questionnaire sexual health and sexual dysfunctions, and the measurement of drug consumption.

ELIGIBILITY:
Inclusion Criteria:

* Crampy pain in the lower abdomen or lumbo-pelvic area between 8 hours and 4 days after menstrual bleeding.
* Clinical evolution of at least three menstrual cycles with said pathology.
* Moderate menstrual pain or severe intensity, minimum 5 VAS scale.
* Regular menstrual cycle, between 21 and 35 days.
* Accept informed consent.

Exclusion Criteria:

* Being receiving any other physiotherapeutic or pharmacological treatment for primary dysmenorrhea during the 3 weeks prior to the beginning of the intervention.
* Suffering from cardiovascular diseases, prolapse, amenorrhea, hemophilia, tumor or infectious processes, use of IUDs, consumption of oral contraceptives or suffering from any injury that affects the sensory-motor function.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Visual Analogue Scale (pain) during menstruation at week 4, 8 and 10. | Baseline and week 4, 8 and 10
  Measured before the treatment in each meeting, asking about the pain during the last menstrual period. The higher is the value of the scale, the worse.
Change from Baseline in the Specific Quality of Life Questionnaire Related to Menstruation CVM-22 at weeks 4, 8 and 10 | Baseline and weeks 4, 8 and 10
  The CVM-22, self-administered Likert type, is made up of 22 items. The questionnaire score ranges from 0 to 66, where the higher the score the worse the CVM-22.
Change from Baseline in the Questionnaire on sexual health and detection of female sexual dysfunctions in primary care (SyDSF-AP) at weeks 4, 8 and 10 | Baseline and weeks 4, 8 and 10
  Self-administered questionnaire of 20 closed questions, although 8, 9 and 19 have an open component, and 1 is an open question, which is integrated into domains. Those of the descriptive sociodemographic domain and the health condition help to know the profile of the surveyed women, as well as the factors that may influence their sexuality. The domain of sexual function ranges from question 10 to 18 and is answered using a Likert scale of 5 values. In addition, question 20 has been included to assess satisfaction with your partner from 0 to 10. Finally, question 21 is open to collect the comments that may arise during the completion of the questionnaire.
change from baseline in the values of the pressure algometer measured on 9 different points at weeks 4, 8 and 10. | Pre-intervention and post-intervention in Baseline and weeks 4 and 8. Another measure without intervention in week 10.
  The Pressure Threshold is defined as the minimum pressure that triggers a painful response. The WAGNER brand "FORCE TEN" pressure algometer was used to quantify the Pressure Thereshold at the 9 sensitive pressure points of dysmenorrhea. The rubber tip was used to focus the pressure exerted by the evaluator and it was placed perpendicular to each point. The measurements were carried out 3 times for each point (with 10 seconds of difference between each measurement, 30 before moving on to another point) and calculating the mean value. Before carrying out the measurements, the patients were instructed in the procedure, giving as an example an area not included in the assessment. When the pressure sensation started to be painful, they should tell the evaluator.
Change from baseline in Medication intake during the menstrual period at weeks 4, 8 and 10. | Baseline and weeks 4, 8 and 10
  The average consumption of NSAIDs by the dose of medication used, self-reported responses by the participants. It will be recorded in a journal that will be given to them to write down.

CONTACTS AND LOCATIONS:
Overall Officials: François Ricard, DO, Study Director — Escuela Osteopatía Madrid
Locations (1):
- Miriam Corona Lozano, Arcos de la Frontera, Cádiz, Spain